CLINICAL TRIAL: NCT05786755
Title: Compositional Shift of Gut Microbiome According to the Complications in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Liver cirrhosis, gut microbime
Record Dates: First submitted 2023-02-06; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Healthy Control: Total number of 52 Healthy Control Included in the study
- Alcoholic Control: Total number of 46 Alcoholic Control Included in the study
- Only Cirrhosis: Total 10 patients with only cirrhosis (n= 10, age 66.66±13.51 years) are included in this study
- Cirrhosis+ HCC: Total 26 patients with Cirrhosis+ hepatocellular carcinoma (HCC) (n= 26, age 61.61±9.85 years) are included in this study
- Cirrhosis+ Varices: Total 7 patients with Cirrhosis+ Varices (n= 7, age 48.42±15.80 years) are included in this study
- Cirrhosis+ Ascites: Total number of 26 patients with Cirrhosis+ Ascites (n= 26, age 55.96±8.51years) are included in this study
- Cirrhosis+ 2 Complications: Total number of 44 patients with cirrhosis with 2 complications (n=44, age 57.84±9.18 years) are included in this study
- Cirrhosis+ 3 Complications: Total number of 29 patients with cirrhosis and 3 or more complication (n=29, aged 59.64±12.61 years) are included in this study

SUMMARY:
Change in gut microbiome is closely associated with liver cirrhosis diseases initiation, progression, establishment, and severity. Nevertheless, compositional alterations in gut microbiome during cirrhosis development still not been evaluated, comprehensively. Here, investigators compared the gut microbial composition in cirrhosis patients to encompassing the gut microbial role in whole spectrum of disease.

DETAILED DESCRIPTION:
Stool samples were collected prospectively from 240 participants (Healthy Control (HC=52) + Alcoholic Control (HC=46) + cirrhosis patients (n=142)). 16S rRNA (ribosomal ribonucleic acid) gene sequencing were performed using the MiSeq sequencer on the illumine platform and based on the phylogenetic relationship,16S-based Microbiome Taxonomic Profiling was performed to discovery gut microbial compositional shift along with cirrhosis severity progression.

ELIGIBILITY:
Inclusion Criteria:

1. Registered in the Hallym University Hospital
2. Presented initially sign of liver cirrhosis
3. Patients must have the following laboratory parameters at screening:

   1. Alanine aminotransferase (ALT) ≤10 × upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST) ≤10 × ULN
   3. Hemoglobin ≥12 g/dL for male, ≥11 g/dL for female patients
   4. Platelets ≥ 50,000/mm3
   5. International normalized ratio (INR) ≤1.5 × ULN unless patient has known haemophilia or is stable on an anticoagulant regimen affecting INR.
   6. Albumin ≥3g/dL.
   7. Direct bilirubin ≤1.5 × ULN h) HbA1c ≤10.0%

   i) Creatinine clearance (CLcr) ≥60 mL/min, as calculated by the Cockcroft-Gault equation.

   -

   Exclusion Criteria:
   * Pregnant Female

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Microbiome Taxonomic Profiling was performed on 240 stool samples (Healthy Control (HC=52) + Alcoholic Control (HC=46) + cirrhosis patients (n=142)). All 142 patients were classified in six groups based on compilation: only cirrhosis, cirrhosis with hepatocellular carcinoma (HCC), cirrhosis with varices, cirrhosis with ascites, cirrhosis with 2 complications and cirrhosis with 3 or more complication.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Gut microbial compositional signature in liver cirrhosis and liver cirrhosis complications. | 2 years
  Gut microbial biomarkers, such as bacterial DNA and metabolic products in the feces, can provide valuable information about the gut microbiome in patients with decompensated cirrhosis, and may be useful in predicting the risk of complications and monitoring disease progression. However, more research is needed to fully understand the role of gut microbiota in decompensated cirrhosis and its complications, and to determine the utility of gut microbial biomarkers as a diagnostic or therapeutic tool in liver cirrhosis and cirrhosis with complications. Therefore, in this clinical trial the investigator will identify cirrhosis dependent bacterial species and metabolites which can have the ability to replace the invasive clinical biomarker for early detection of decompensation in cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Suk, PhD, Principal Investigator — Chuncheon Sacred Hallym hospital
Locations (1):
- Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No